CLINICAL TRIAL: NCT04835051
Title: Implementation Research on an Urban Private Sector Model of IYCF Counseling in Private Health Facilities in Lagos State
Brief Title: Alive & Thrive Nigeria Breastfeeding Promotion in Urban Private Facilities Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20576
Record Dates: First submitted 2021-02-23; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-01

CONDITIONS: Breastfeeding
Keywords: Exclusive breastfeeding; Early initiation of breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding promotion (Other): The breastfeeding promotion intervention included training for health workers, interpersonal communication (in person and digital) between providers and pregnant/breastfeeding women, and mass media.
  Interventions: Behavioral: Breastfeeding promotion
- Comparison (No Intervention)

INTERVENTIONS:
Behavioral: Breastfeeding promotion — The intervention included training of health workers in private health facilities to provide in-person breastfeeding counseling to pregnant women and women with a child <6 months during clinic visits. The health workers also offered a mobile phone support component for appointment reminders, breastfeeding SMS and WhatsApp messages, WhatsApp breastfeeding support groups, informational materials (posters and foldable pocket-sized cards), and family engagement activities. Breastfeeding-related mass media through television and radio spots was available state-wide, including to women in intervention and comparison facilities.
  Arms: Breastfeeding promotion

SUMMARY:
The purpose of this study was to evaluate the effect of a breastfeeding promotion intervention on breastfeeding intentions, early initiation of breastfeeding, and exclusive breastfeeding among clients in private health facilities in Lagos, Nigeria.

DETAILED DESCRIPTION:
This was a longitudinal cohort study designed to evaluate and measure the implementation processes of a breastfeeding counseling and support intervention offered to pregnant and postpartum women in private health facilities in Lagos State, Nigeria. This study was conducted as part of the Alive & Thrive Nigeria program, implemented by FHI 360 and partners. RTI led the design, implementation, and analysis for the study, with Datametrics Associates Ltd. serving as the data collection partner in Nigeria. The study took place in 20 private health facilities. Ten facilities were assigned to intervention and 10 to comparison based on their location within the existing intervention and comparison local government areas (LGAs) for our overall impact evaluation of the Alive & Thrive program in Nigeria (NCT02975063). To be included in the study, facilities had to provide maternity and pediatric services, such as antenatal care, postnatal care, and immunizations, and be registered with the Association of General and Private Medical Practitioners of Nigeria and the Health Facility Monitoring and Accreditation Agency. To ensure that the investigators would achieve their sample size, selected facilities with a monthly average of ≥40 antenatal clients and ≥20 deliveries over 3 months. All eligible women attending antenatal care on the days of data collection were invited to participate until the target enrollment at each facility was achieved. The investigators collected survey data from a cohort of 1,200 women (600 per study arm) during the third trimester of pregnancy and when their child was 6 weeks and 24 weeks. The purpose of the surveys were to obtain data on the women's breastfeeding intentions (third trimester) and practices (6 weeks and 24 weeks), their breastfeeding knowledge and attitudes, and their exposure to the intervention. To measure implementation outcomes, the investigators conducted 180 observations of client-provider interactions among a subset of women enrolled in the study and then completed a short exit interview with the women immediately after their facility visit. In addition, the investigators conducted qualitative interviews with 20 health providers and facility managers/owners in the intervention facilities at the end of the intervention to learn about the facilitators and barriers to implementation.

ELIGIBILITY:
Inclusion:

* Women ≥18 years old, third trimester
* Current Client of a private health facility
* Infant alive at 6 and 24 weeks postpartum

Exclusion:

* Infant died
* Infant unable to breastfeed

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1220 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding | 6 weeks
  The proportion of infants exclusively breastfed on the previous day
Exclusive breastfeeding | 24 weeks
  The proportion of infants exclusively breastfed on the previous day

SECONDARY OUTCOMES:
Early initiation of breastfeeding | At birth
  The proportion of infants who started breastfeeding within 1 hour of birth

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Flax, PhD, Principal Investigator — RTI International
Locations (20):
- Nigeria (20):
  - Albina Majeed Clinic, Lagos
  - Ayodele Medical Centre, Lagos
  - Crystal Specialist, Lagos
  - Edmac Medical Centre, Lagos
  - Eko Hospital, Lagos
  - El-Dunamis Medical Centre, Lagos
  - Faith City Hospital, Lagos
  - Fuja Medical Centre, Lagos
  - Ilogbo Central Hospital, Lagos
  - Isalu Hospital, Lagos
  - Matador Hospital, Lagos
  - Mobonike Hospital, Lagos
  - Modupeoluwa Mat.Home, Lagos
  - Promise Medical Centre, Lagos
  - R-Jolard Hospital, Lagos
  - Rccg Ebute Metta, Lagos
  - Rccg Oke Suna, Lagos
  - Redeemed Maternity Amuwo, Lagos
  - Regina Mundi Catholic Hospital, Lagos
  - Uwemdimo Hospital, Lagos

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared publicly through Harvard Dataverse.
Time Frame: January 31, 2022
Access Criteria: open

REFERENCES:
- [Derived] Flax VL, Ipadeola A, Schnefke CH, Ralph-Opara U, Adeola O, Edwards S, Bose S, Brower AO. Breastfeeding Interpersonal Communication, Mobile Phone Support, and Mass Media Messaging Increase Exclusive Breastfeeding at 6 and 24 Weeks Among Clients of Private Health Facilities in Lagos, Nigeria. J Nutr. 2022 May 5;152(5):1316-1326. doi: 10.1093/jn/nxab450. PMID 35015869